CLINICAL TRIAL: NCT00955708
Title: Condition of Approval Study: Longitudinal Surveillance Registry of the ACUITY Spiral Lead
Brief Title: Longitudinal Surveillance Registry (LSR) of ACUITY Spiral
Status: Terminated | Type: Observational
Why Stopped: Early termination was granted by FDA based on study results meeting the post approval requirements.
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: LSR of ACUITY Spiral
Record Dates: First submitted 2009-08-04; First posted 2009-08-10 (Estimated); Results first posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Implants: Patients successfully implanted with the ACUITY Spiral Lead
  Interventions: Device: ACUITY Spiral Left Ventricular Lead

INTERVENTIONS:
Device: ACUITY Spiral Left Ventricular Lead — The implant of the ACUITY Spiral Lead

SUMMARY:
The primary purpose of the LSR of ACUITY Spiral is to evaluate and report on the long-term performance of the ACUITY Spiral Left Ventricular Lead.

ELIGIBILITY:
Inclusion Criteria:

* Has been or will be implanted with the ACUITY Spiral Lead within 29 days
* Plans to remain in the long-term care of his/her enrolling physician
* Is willing and capable (or appropriate legal representative) of authorizing access to and use of health information as required by an institution's institutional review board (IRB)
* Is willing and capable (or appropriate legal representative) of providing authorization for participation in the registry

Exclusion Criteria:

* Is unable or unwilling to comply with the protocol requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population will be a broad base representative of those recieving the ACUITY Spiral lead.
Sampling Method: Non-Probability Sample
Enrollment: 1308 (Actual)
Dates: Start 2009-08-04 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Hedrich, MD, Study Director — Boston Scientific Corporation
Locations (97):
- United States (97):
  - Birmingham Heart Clinic, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Tri-City Cardiology, Mesa, Arizona
  - Arizona Arrhythmia Research Center, Scottsdale, Arizona
  - Pima Heart Physicians, Tucson, Arizona
  - Cardiology Associates of Northeast Arkansas, Jonesboro, Arkansas
  - Heart Clinic Arkansas, Little Rock, Arkansas
  - Comprehensive Cardiovascular Medical Group, Bakersfield, California
  - Belott Cardiology, El Cajon, California
  - Fullerton Cardiovascular, Fullerton, California
  - Cardiac Device Rhythm Specialists, Los Angeles, California
  - Cedars - Sinai Medical Center, Los Angeles, California
  - Memorial Hospital, Modesto, California
  - Cardiac Rhythm Specialists, Inc., Northridge, California
  - Cardiovascular Consultants, Oakland, California
  - Orange County Heart Institute, Orange, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Truong D Duong Cardiac Electrophysiology, Riverside, California
  - Regional Cardiology Associates, Sacramento, California
  - Sansum Clinic, Santa Barbara, California
  - Bethesda Memorial Hospital, Atlantis, Florida
  - Heart and Vascular Institute of Florida, Clearwater, Florida
  - Miami International Cardiology Consultants, Miami, Florida
  - Complete Cardiology Care, New Smyrna Beach, Florida
  - Orlando Regional Hospital, Orlando, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - West Coast Arrhythmia Center, Trinity, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Medical College of Georgia Health, Augusta, Georgia
  - Northeast Georgia Heart Center, Gainesville, Georgia
  - Georgia Arrhythmia Consultants, Macon, Georgia
  - St Lukes Idaho Cardiology Assoc., Boise, Idaho
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Heart Care Research Foundation, Mokena, Illinois
  - Northern Indiana Research Alliance, Fort Wayne, Indiana
  - St. Mary Medical Center - Indiana, Hobart, Indiana
  - Via-Christi Regional Medical Center, Wichita, Kansas
  - Southern Kentucky Heart Institute, Bowling Green, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - St. Joseph Hospital, Lexington, Kentucky
  - Commonwealth Cardiology, Louisville, Kentucky
  - Baltimore Heart Association, Randallstown, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Steward St. Elizabeth's Medical Center, Boston, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Heart Care, Detroit, Michigan
  - Cardiology Consultants of East Michigan, Flint, Michigan
  - West Michigan Heart, Grand Rapids, Michigan
  - Providence Hospital, Southfield, Michigan
  - St. Mary's Duluth Clinic, Duluth, Minnesota
  - Missouri Heart Center, Columbia, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Cox Health, Springfield, Missouri
  - Metro Heart Group South County, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - New Jersey Cardiology Associates, West Orange, New Jersey
  - Capital Cardiology Associates, Albany, New York
  - Island Cardiac Specialists, Garden City, New York
  - Columbia University Medical Center, New York, New York
  - Mid-Carolina Cardiology, Charlotte, North Carolina
  - Pinehurst Cardiology Consultants, Pinehurst, North Carolina
  - Christ Hospital - Cincinnati, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Regional Cardiovascular Medical Center, Steubenville, Ohio
  - Genesis Healthcare System, Zanesville, Ohio
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Associated Cardiologists, Harrisburg, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Cardiovascular Associates of Rhode Island, Providence, Rhode Island
  - Columbia Cardiology, Columbia, South Carolina
  - PeeDee Cardiology Associates, Florence, South Carolina
  - Heart Doctors, Rapid City, South Dakota
  - Memphis Heart Clinic, Memphis, Tennessee
  - Amarillo Heart Group, Amarillo, Texas
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - Heart Hospital of Austin, Austin, Texas
  - Cardiology Care Consultants, El Paso, Texas
  - Hall Garcia Cardiology, Houston, Texas
  - Houston Electrophysiology Associates, Houston, Texas
  - Willowbrook Cardiovascular Associates, Houston, Texas
  - EP Heart, The Woodlands, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - Intermountain Medical Center, Murray, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Virginia Heart, Falls Church, Virginia
  - Richmond Cardiology Associates, Mechanicsville, Virginia
  - Overlake Medical Center, Bellevue, Washington
  - St. Joseph Hospital, Bellingham, Washington
  - Swedish Medical Center, Seattle, Washington
  - Heart Clinics Northwest, Spokane, Washington
  - Wheaton Franciscan Healthcare, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Implants: Patients successfully implanted or underwent an attempted implant with the ACUITY Spiral Lead
  ACUITY Spiral Left Ventricular Lead: The implant of the ACUITY Spiral Lead
Period: Overall Study
Arm/Group | Implants
Started | 1308
Completed | 250
Not Completed | 1058
Not completed — Death | 269
Not completed — Lost to Follow-up | 72
Not completed — Physician Decision | 36
Not completed — Protocol Violation | 134
Not completed — Registry Conclusion | 186
Not completed — Product removed from service | 94
Not completed — Patient Refused to participate further | 116
Not completed — Closure of study location | 60
Not completed — Patient changed care provider/moved | 91

BASELINE CHARACTERISTICS:
Population: Baseline data includes data on the patients that received an implant or underwent an attempted implant. This does not include intent patients who were consented but did not participate in the trial and did not undergo anesthesia.
Arm/Group | Implants
Number analyzed (Participants) | 1303
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 387
  >=65 years | 916
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 357
  Male | 946
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 16
  Native Hawaiian or Pacific Islander | 5
  Black or African American | 124
  White | 1065
  Bosnian | 1
  East Indian | 1
  Filipino | 1
  Middle Eastern | 1
  Russian | 1
  Unknown | 29
  Hispanic or Latino | 52
  Vietnamese | 1
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 2
  United States | 1301
QRS Duration [Mean (Standard Deviation); unit: Milliseconds] — Population: QRS Duration value unavailable for 49 subjects
  Milliseconds
    number analyzed (Participants) | 1254
    (all) | 150 (31)
PR Interval [Mean (Standard Deviation); unit: milliseconds] — Population: PR Interval (ms) unavailable for 354 subjects
  milliseconds
    number analyzed (Participants) | 958
    (all) | 183 (55)
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: percentage] — Population: Left Ventricular Ejection Fraction unavailable for 25 subjects
  percentage
    number analyzed (Participants) | 1278
    (all) | 26.8 (7.9)
Arrhythmia Conduction Disorder [Count of Participants; unit: Participants] — Population: Arrhythmia Conduction Disorder was unavailable for 23 subjects
  Participants
    number analyzed (Participants) | 1285
    Left Bundle Branch Block | 691
    Right Bundle Branch Block | 149
    Nonspecific Intraventricular Delay | 228
    No Arrhythmia Conduction Disorder | 140
    Unknown | 77

OUTCOME MEASURES:

1. Primary Outcome: Chronic Left Ventricular Lead-related Complication Free Rate
Time Frame: Date of enrollment to study completion (Date of 5 year follow-up, withdrawal or death).
Measure: Number (95% Confidence Interval); unit: Percent free from event
Arm/Group | Implants
Number analyzed (Participants) | 1303
Percent free from event | 95.3 [94.0 to NA] — Interval is only calculated for the lower end. The method is defined as the lower one-sided 95% confidence interval compared to the confidence boundary of 92.5%.
Statistical Analysis 1: Comparison: Implants; The endpoint data reflected here is a modified primary endpoint analysis requested by the Food and Drug Administration early in the registry to include data that is related to the left ventricular lead function in a chronic setting; Test type: Other — Primary endpoint was estimated using the Kaplan-Meier method. In addition, Greenwood's formula was used to calculate the lower one-sided 95% confidence bound; Kaplan-Meier Rate = 95.3, 95.0% CI 1-sided [lower limit 94.0] — The lower one-sided 95% confidence bound was pre-specified to be greater than 92.5%
Statistical Analysis 2: Comparison: Implants; The non-modified primary endpoint analysis initially included confirmed chronic LV lead related complications that result in permanent loss of therapy, invasive intervention, injury or death, and are deemed attributable to a structural lead failure by an independent Clinical Events Committee (CEC). These results are represented here; Test type: Other — [test comment as in outcome 1, analysis 1]; Kaplan-Meier Rate = 100, 95% CI 1-sided [lower limit 100]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of enrollment into the trial through completion of the registry at 5 years, date of withdrawal or death.
Description: Adverse event reporting for the LSR of ACUITY Spiral trial included all pulse generator, or lead (Left Ventricular, Right Ventricular or atrial leads are all included) related events occurring at or after implant. Reportable events are defined as inappropriate performance of the pulse generator or leads that result in an undesirable or unanticipated procedure or clinical occurrence.
Arm/Group | Implants
All-Cause Mortality (participants affected / at risk) | 269/1303
Serious Adverse Events (participants affected / at risk) | 117/1303
Other Adverse Events (participants affected / at risk) | 131/1303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implants (N=1303)
Extracardiac Stimulation, Left Ventricular (Cardiac disorders) | 10 (10)
Lead Dislodgment, Left Ventricular (Cardiac disorders) | 29 (29)
Threshold Related, Left Ventricular (Cardiac disorders) | 19 (19)
Ventricular Tachycardia (Cardiac disorders) | 2 (2)
Cardiac Vessel Dissection (Surgical and medical procedures) | 1 (1)
Lead Revision for no heart failure improvement, Left Ventricular (Surgical and medical procedures) | 1 (1)
Accelerated Ventricular Rhythm (Cardiac disorders) | 2 (2)
Atrial Arrhythmia (Cardiac disorders) | 1 (1)
Pulse Generator Possible Malfunction (Product Issues) | 2 (2)
Pulse Generator Related (Surgical and medical procedures) | 1 (1) — Lead to device connection re-evaluated
Erosion/Migration (Surgical and medical procedures) | 9 (10)
Heart Failure Decompensation (Cardiac disorders) | 2 (2)
Hematoma (Blood and lymphatic system disorders) | 2 (2)
Inability to provide therapy, pulse generator (Surgical and medical procedures) | 5 (5)
Infection, Procedure related (Surgical and medical procedures) | 10 (10)
Pneumothorax (Injury, poisoning and procedural complications) | 1 (1)
Premature Ventricular Contractions (PVCs) (Cardiac disorders) | 1 (1)
Impedance Related, Atrial Lead (Cardiac disorders) | 1 (1)
Infection, Atrial Lead (Injury, poisoning and procedural complications) | 1 (1)
Lead Dislodgment, Atrial Lead (Cardiac disorders) | 6 (6)
Sensing Related, Atrial Lead (Cardiac disorders) | 1 (1)
Threshold Related, Atrial Lead (Cardiac disorders) | 2 (2)
Cardiac Perforation, Right Ventricular (Surgical and medical procedures) | 1 (1)
Impedance Related, Right Ventricular (Cardiac disorders) | 3 (3)
Inappropriate Tachy Therapy, Right Ventricular (Cardiac disorders) | 3 (3)
Infection, Right Ventricular (Injury, poisoning and procedural complications) | 1 (1)
Lead Dislodgment, Right Ventricular (Surgical and medical procedures) | 5 (5)
Pneumothorax, Right Ventricular (Injury, poisoning and procedural complications) | 1 (1)
Sensing Related, Right Ventricular (Cardiac disorders) | 1 (1)
Threshold Related, Right Ventricular (Cardiac disorders) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implants (N=1303)
Extracardiac Stimulation, Left Ventricular (Cardiac disorders) | 77 (88)
Threshold Related, Left Ventricular (Cardiac disorders) | 26 (33)
Inappropriate Tachy Therapy, Pulse Generator (Cardiac disorders) | 28 (36)

LIMITATIONS AND CAVEATS:
Early termination was granted based on study results. The study was one-armed observational. The expected performance / safety of left ventricular leads has been established; permitting comparison to a pre-defined performance standard.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-12-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT00955708/Prot_000.pdf
  • Statistical Analysis Plan (2013-07-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT00955708/SAP_001.pdf